CLINICAL TRIAL: NCT04949815
Title: Case Series; Awake Craniotomy for Brain Arteriovenous Malformation - Experience From a Tertiary Care Center in a Low- And Middle-Income Country
Brief Title: Awake Craniotomy for Arteriovenous Malformation
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, S Ather Enam, MD PhD, Professor, Aga Khan University
Other Study IDs: 2019-1436-4508
Record Dates: First submitted 2021-06-23; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Awareness, Anesthesia; Arteriovenous Malformations
MeSH Terms: conditions — Intraoperative Awareness; Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aimed to retrospectively review cases of brain arteriovenous malformation that were surgical resected with the patient awake during the procedure.

DETAILED DESCRIPTION:
Four patients' charts were retrospectively reviewed and neurological status before and after awake craniotomy was assessed to look for any deterioration.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of arteriovenous malformation in brain
* Awake craniotomy for surgical resection of arteriovenous malformation

Exclusion Criteria:

* Patients with incomplete records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients, irrespective of age and gender, who underwent awake craniotomy under scalp block for resection of brain AVMs at our hospital were reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Change in neurological status after surgery including GCS, cranial nerve functions and motor power in all four limbs (according to MRC scale). | 10 days
  Comparison of pre-operative and post-operative neurological status to assess whether there was net improvement or deterioration. Pre-operative neurological status was assessed at the time of hospital admission and post-operative neurological status was assessed after 10 days of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan